CLINICAL TRIAL: NCT04803812
Title: Supporting the Wellness of Ontario Physicians During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Medical Association (Other)
Collaborators: The Behavioural Insights Team (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 39707
Record Dates: First submitted 2021-02-08; First posted 2021-03-18 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Mental Health Wellness 1; Anxiety; Happiness
MeSH Terms: conditions — Anxiety Disorders | interventions — Parturition

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Receive weekly SMS containing wellness stories shared by other Ontario physicians (Experimental)
  Interventions: Other: Remote SMS (short message service, also known as "text message") delivery
- Receive weekly SMS containing aim wellness resources/strategies. (Experimental)
  Interventions: Other: Remote SMS (short message service, also known as "text message") delivery
- Receive weekly SMS combining wellness stories & resources/strategies (Experimental)
  Interventions: Other: Remote SMS (short message service, also known as "text message") delivery

INTERVENTIONS:
Other: Remote SMS (short message service, also known as "text message") delivery — Assessing the comparative effects of SMS types (storytelling; resources/strategies; and a combination of both) on physician wellbeing.

SUMMARY:
In light of the coronavirus pandemic, the challenge of physician burnout has taken on a new urgency. Long-hours and difficult, sometimes unsafe work conditions are creating a severe strain for emergency physicians and others on the frontlines of Ontario's response to COVID-19. There are a variety of evidence-informed ways that physicians can protect their wellbeing with modest investments of time and energy that will be applied. The evaluation will be a randomized trial comparing the outcomes from each of the three treatment arms. Researchers may also use a pre-post comparison with control parameters to conduct an exploratory analysis to assess efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Active membership to the Ontario Medical Association (OMA). Up-to-date cell phone information registered to the OMA.

Exclusion Criteria:

* Participation in the OMA Physician Burnout Task Force. Opt-out from the intervention.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19124 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Wellbeing (Short Warwick-Edinburgh Mental Well-being Scale measure) | 6 months
  Self-reported wellbeing scores, as measured by the short Warwick-Edinburgh Mental Well-being Scale--(S)WEMWBS. The (S)WEMWBS is designed to measure positive mental wellbeing and asks people to what extent they agree with statements such as "I've been feeling optimistic about the future", "I've been feeling relaxed", and "I've been feeling close to people". This scale has a range of 7 to 35; higher scores indicate higher positive mental wellbeing.

SECONDARY OUTCOMES:
Happiness (UK ONS measure) | 6 months
  Self-reported happiness scores, as measured through weekly pulse surveys using a question developed by the UK Office for National Statistics (ONS) - hereby referred to as ONS-happiness ("on a scale where 0 is "not at all" and 10 is "completely", overall, how happy did you feel yesterday?"). This scale has a range from 0 to 10, with higher scores indicating greater happiness.
Anxiety (UK ONS measure) | 6 months
  Self-reported anxiety scores, as measured through pulse surveys using an ONS question, hereby referred to as ONS-anxiety ("on a scale where 0 is "not at all" and 10 is "completely", overall, how anxious did you feel yesterday?"). This scale has a range from 0 to 10, with higher scores indicating greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: James Wright, Principal Investigator — Ontario Medical Association
Locations (1):
- Ontario Medical Association, Toronto, Ontario, Canada